CLINICAL TRIAL: NCT04427930
Title: Long-Term Safety and Efficacy Extension Study Of Autologous Adipose-Derived Mesenchymal Stem Cells 『JOINTSTEM』 in Patients With Knee Osteoarthiritis: A Phase III Extension Study
Brief Title: Follow-up Study for Participants of Jointstem Phase 3 Clinical Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSR-CTph3-JS1_FU
Record Dates: First submitted 2020-05-20; First posted 2020-06-11 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JOINTSTEM (Experimental): Long Term Follow-up after Jointstem Transplantation
  Interventions: Biological: JOINTSTEM

INTERVENTIONS:
Biological: JOINTSTEM — Autologous Adipose Tissue derived MSCs

SUMMARY:
The purpose of this follow-up study is to investigate the efficacy and safety of autologous Adipose Tissue derived Mesenchymal stem cells (JOINTSTEM®) in patient with severe Knee Osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Participants of Jointstem Phase 3 Clinical Trial
* Participates who signed informed consent document of this study

Exclusion Criteria:

* No applicable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 5 Years
  Incidence of adverse events from baseline to 5 Years

SECONDARY OUTCOMES:
Change of Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) scores from baseline | 5 Years
  Pain, stiffness, and physical function of the knee will be measured by the WOMAC score
WOMAC 3 subscale score | 5 Years
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities (WOMAC)
SF-36 | 5 Years
  The SF(Short Form)-36 Health Survey is a 36-item, patient-reported survey of patient health.
Measuring of Kellgren-Lawrence grade | 1, 2, 3, 4, 5 Years
  Measuring of Kellgren-Lawrence grade through X-ray
Measuring of Femoro-tibial anatomical angle(FTA) | 1, 2, 3, 4, 5 Years
  Measuring of FTA through X-ray
Measuring of Hip-Knee-Ankle angle(HKA) | 1, 2, 3, 4, 5 Years
  Measureing of HKA through X-ray
Measuring of Joint Space Width | 1, 2, 3, 4, 5 Years
  measuring Joint Space Width through X-ray
MRI scan | 1, 2, 3, 4, 5 Years
  The cartilage defect area is measured using MRI

CONTACTS AND LOCATIONS:
Overall Officials: KANGIL KIM, Principal Investigator — KyungHee University Gangdong Hospital; WOOSUK LEE, Principal Investigator — Gangnam Severance Hospital; KICHEOR BAE, Principal Investigator — Keimyung University Dongsan Medical Center; YONG IN, Principal Investigator — The Catholic University of Korea
Locations (4):
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - KyungHee University Gangdong Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul